CLINICAL TRIAL: NCT03670628
Title: Randomized Control Trial of Low Intensity Shockwaves for the Treatment of Erectile Dysfunction. 12- Month Follow-Up of a Double-Blinded, Sham-Controlled Study.
Brief Title: Low Intensity Shockwaves Therapy for the Treatment of Erectile Dysfunction. 12- Month Follow-Up
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Due to COVID-19 Pandemic
Sponsor: University of Miami (Other)
Responsible Party: Principal Investigator, Ranjith Ramasamy, MD, Director of Male Fertility/ Andrology department, University of Miami
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 20180651; 20181840 (Other: western IRB)
Record Dates: First submitted 2018-09-10; First posted 2018-09-13 (Actual); Results first posted 2023-07-10 (Actual); Last update posted 2023-07-10 (Actual); Status verified 2023-06

CONDITIONS: Erectile Dysfunction
MeSH Terms: conditions — Erectile Dysfunction | interventions — Extracorporeal Shockwave Therapy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- 720 shockwave therapy Group (Active Comparator): Participants in this group will receive a total of 5 daily sessions of shockwave therapy within a week. Each therapy session will consist of 720 shockwave therapy applied to the penis and to the left and right crus (shaft near the base)
  Interventions: Device: Shockwave therapy
- Sham shockwave therapy (Sham Comparator): Participants in this group will receive a total of 5 daily sessions of sham shockwave therapy within a week. Sham therapy will be applied to the penis and to the left and right crus (shaft near the base).
  Interventions: Other: Sham shockwave therapy

INTERVENTIONS:
Device: Shockwave therapy — Each therapy session, lasting about 20 minutes, will deliver 720 shockwave therapy applied to the penis and to the left and right crus (shaft near the base)
  Arms: 720 shockwave therapy Group
Other: Sham shockwave therapy — Each therapy session, lasting about 20 minutes, will deliver sham shockwave therapy applied to the penis and to the left and right crus (shaft near the base)
  Arms: Sham shockwave therapy

SUMMARY:
The purpose of this study is to evaluate the safety and effectiveness of the shockwave therapy to treat Erectile Dysfunction.

ELIGIBILITY:
Inclusion Criteria:

* The patient must be able willing and able to provide informed consent.
* The patient is a male between 30 and 70 years of age (inclusive).
* The patient has erectile dysfunction (ED) based of IIEF scores.
* The patient has been in a stable relationship for over 3 months prior to enrollment.
* A minimum of 2 sexual attempts per month for at least one month prior to enrollment - as documented by International Index of Erectile Dysfunction (IIEF)
* The patient is suffering from erectile dysfunction lasting for over 6 months and not more than 5 years as per history provided by patient.
* IIEF-EF score between 16 and 25.
* Testosterone level 300-1000 ng/dL within 1 month prior to enrollment. A1C level ≤ 7% within 1 month prior to enrollment

Exclusion Criteria:

* The patient is currently or has participated in another study within the past three months that may interfere with the results or conclusions of this study.
* The patient is under judicial protection (prison or custody).
* The patient is an adult under guardianship.
* The patient refuses to sign the consent.
* History of radical prostatectomy or extensive pelvic surgery.
* Evidence of venous leak.
* Past radiation therapy of the pelvic region within 12 months prior to enrollment.
* Recovering from any cancer within 12 months prior to enrollment.
* Neurological disease such as Alzheimers or Parkinson's disease which affects erectile function at the discretion of the investigator.
* Psychiatric diagnosis or medications such as antidepressants, anxiolytic, antipsychotic that affects erectile function or any other medications at the discretion of the investigator.
* Anatomical malformation of the penis, including Peyronie's disease.
* Testosterone level <300 or >1000 ng/dL within 1 month prior to enrollment.
* A1C level > 7% within 1 month prior to enrollment or history of Insulin dependent diabetes.
* The patient is taking blood thinners and has an international normalized ratio >3.
* Received shockwave treatment at least 6 months before enrollment.

Ages: 30 Years to 70 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2019-05-01 (Actual); Primary Completion 2021-11-12 (Actual); Study Completion 2021-11-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ranjith Ramasamy, MD, Principal Investigator — University of Miami
Locations (1):
- University of Miami, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Unable to complete target enrollment due to COVID-19 pandemic restrictions.
Period: Baseline Visit
Arm/Group | 720 Shockwave Therapy Group | Sham Shockwave Therapy
Started | 13 | 10
Completed | 13 | 10
Not Completed | 0 | 0
Period: Weekly Therapy Sessions
Arm/Group | 720 Shockwave Therapy Group | Sham Shockwave Therapy
Started | 13 | 10
Completed | 5 | 7
Not Completed | 8 | 3
Not completed — Enrollment was halted; participants were unable to attend study visits due to COVID-19 restrictions. | 8 | 3
Period: Month 1 Visit
Arm/Group | 720 Shockwave Therapy Group | Sham Shockwave Therapy
Started | 5 | 7
Completed | 5 | 7
Not Completed | 0 | 0
Period: Waiting Period
Arm/Group | 720 Shockwave Therapy Group | Sham Shockwave Therapy
Started | 5 | 7
Completed | 1 | 1
Not Completed | 4 | 6
Not completed — Enrollment was halted; participants were unable to attend study visits due to COVID-19 restrictions. | 4 | 6
Period: Month 3 Visit
Arm/Group | 720 Shockwave Therapy Group | Sham Shockwave Therapy
Started | 1 | 1
Completed | 1 | 1
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 720 Shockwave Therapy Group | Sham Shockwave Therapy | Total
Number analyzed (Participants) | 13 | 10 | 23
Age, Continuous [Mean (Standard Deviation); unit: years] | 52.4 (10.5) | 51.2 (8.9) | 51.7 (9.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 13 | 10 | 23
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: International Index of Erectile Function (IIEF) Erectile Function Subdomain (EF) Scores.
Description: The IIEF-EF questionnaire has a total score ranging from 0 - 30 with the higher score indicating better erectile function.
Time Frame: Baseline, Month 1, Month 3, Month 6, Month 9, and Month 12
Population: No statistical analyses have been performed or would be considered scientifically appropriate because actual enrollment fell well below target enrollment. Enrollment terminated early as a result of the COVID-19 pandemic.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | 720 Shockwave Therapy Group | Sham Shockwave Therapy
Number analyzed (Participants) | 13 | 10
score on a scale
  Baseline | 18.8 (2.7) | 19.1 (3.6)
  Month 1: number analyzed (Participants) | 5 | 7
  Month 1 | 18.4 (7.1) | 17 (4.5)
  Month 3: number analyzed (Participants) | 1 | 1
  Month 3 | 18 (NA) — None of the data were analyzed because of insufficient participant numbers and power to draw conclusions. | 26 (NA) — None of the data were analyzed because of insufficient participant numbers and power to draw conclusions.

2. Secondary Outcome: Number of Participants Responding 'Yes' to the Sexual Encounter Profile (SEP) Questionnaire
Description: The SEP consists of two questions: 1) Over the past 4 weeks, were you able to insert your penis into your partner's vagina? and 2) Over the past 4 weeks, did your erection last long enough for you to have successful intercourse? Reported will be the number of participants responding yes to the 2 questions.
Time Frame: Baseline, Month 1, Month 3, Month 6, Month 9, and Month 12
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | 720 Shockwave Therapy Group | Sham Shockwave Therapy
Number analyzed (Participants) | 13 | 10
participants
  Baseline | 7 | 2
  Month 1: number analyzed (Participants) | 5 | 6
  Month 1 | 3 | 2
  Month 3: number analyzed (Participants) | 1 | 1
  Month 3 | 1 | 0

3. Secondary Outcome: Erection Hardness Score (EHS)
Description: EHS has a total score ranging from 0 - 4 with the higher score indicating a better erection hardness
Time Frame: Baseline, Month 1, Month 3, Month 6, Month 9, and Month 12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | 720 Shockwave Therapy Group | Sham Shockwave Therapy
Number analyzed (Participants) | 13 | 10
score on a scale
  Baseline | 2.9 (0.3) | 2.8 (0.6)
  Month 1: number analyzed (Participants) | 5 | 7
  Month 1 | 3.4 (0.5) | 3.1 (0.4)
  Month 3: number analyzed (Participants) | 1 | 1
  Month 3 | 3 (NA) — None of the data were analyzed because of insufficient patient numbers and power to draw conclusions. | 4 (NA) — None of the data were analyzed because of insufficient patient numbers and power to draw conclusions.

ADVERSE EVENTS:
Time Frame: 3 months
Arm/Group | 720 Shockwave Therapy Group | Sham Shockwave Therapy
All-Cause Mortality (participants affected / at risk) | 0/13 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/13 | 0/10
Other Adverse Events (participants affected / at risk) | 0/13 | 0/10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-05-02): https://cdn.clinicaltrials.gov/large-docs/28/NCT03670628/Prot_SAP_000.pdf